CLINICAL TRIAL: NCT03650296
Title: Evaluating Different Pediatric Emergency Rulers in a Manikin Study - How Fast and Correct Are They
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: ePER vs PS vs PNL
Record Dates: First submitted 2018-07-08; First posted 2018-08-28 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Time Until Identification of Defined Parameter

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Resusci Baby: Resusci Baby used for the simulated emergency scenario
  Interventions: Device: ePER vs PS vs PaedER
- MegaCode-Kid: MegaCode-Kid used for the simulated emergency scenario
  Interventions: Device: ePER vs PS vs PaedER
- Ambu® Junior: Ambu® Junior used for the simulated emergency scenario
  Interventions: Device: ePER vs PS vs PaedER

INTERVENTIONS:
Device: ePER vs PS vs PaedER — see detailed description of methods

SUMMARY:
Comparison of three different pediatric emergency rulers for length-based body weight estimation in pediatric emergencies.

Primary outcome is the time needed to identify four defined parameters from the pediatric emergency rulers during a low-fidelity pediatric emergency scenario (cardiac arrest). Secondary outcome is the correctness of the identified parameters and the percentage deviation from the correct value.

DETAILED DESCRIPTION:
Medical team members (consultants, residents and nurses) of the department of Anaesthesia at the University Children's Hospital Zurich were asked to participate in this study. If they were not familiar with one of the three devices written informed consent was obtained and the participant included in this study. This exclusion criteria was necessary to prevent a bias by already knowing where to find the information of interest.

The pediatric emergency rulers investigated were:

The electronic Pediatric Emergency Ruler (ePER) is based on the Continuous Length-based Algorithm for Weight & Age Rating (CLAWAR). This digital algorithm is based on gender-specific Swiss length-weight and Swiss length-age growth charts and uses the 50th percentile to estimate the patient's body weight and age. CLAWAR was recently published and showed a higher accuracy compared to a conventional emergency tape. A smartphone application (APP) was programmed based on CLAWAR and is utilized in the ePER. CLAWAR, the APP and ePER were developed by the department of Anaesthesia at the University Children's Hospital Zurich.

The "Paulino System" (PS; Paulino-System & Altonaer Werbewerkstatt, Hamburg, Germany) utilizes a ruler with 27 length-based weight categories for a body length from 44 to 151 cm. Separate from this ruler weight estimation ruler drug dosing, sizes of medical equipment, and vital parameters for each of the 27 weight categories can be found in a color-coded booklet.

The "Paediatric Emergency Ruler" (PaedER; Alpha 1 Werbedesign e.K., Falkenberg, Germany) is a paediatric emergency tape certified for clinical use in Europe and applicable for patients with a body length between 44 and 140 cm. PaedER is grouped in 11 length based weight categories to assist estimation of patients' body weight, to suggest drug dosing (mg and ml) for the most common emergency drugs and to recommend adequate sizes of medical equipment and norm-values for vital signs. The basic idea is identical to the of the Broselow Luten tape.

All participants were instructed for the use of the three pediatric emergency rulers and were given time to practice with each device using one training manikin (Sim-Baby)

After they felt comfortable using the devices the participants were randomly assigned to use each device only once with one of three different manikins:

* Resusci Baby, Laerdal/Dräger Medical Switzerland AG, Liebefeld, Switzerland
* MegaCode-Kid, Laerdal/Dräger Medical Switzerland AG, Liebefeld, Switzerland
* Ambu® Junior, Ambu® GmbH, Bad Nauheim, Germany

Each manikin was only used once for the same participant. This guaranteed that the participants were blinded for the manikins.

The low-fidelity pediatric emergency scenario simulated was a cardiac arrest and the participants were asked to identify the following information from the pediatric emergency rulers:

* Estimated body weight
* Joule suggested for defibrillation
* Recommended epinephrine dose
* Suggested endotracheal tube size

Participants stood aside from the manikin with a pediatric emergency ruler in their hand. After they stated they were ready, the facilitator started a countdown from three and gave the command to start. This setting was identical for all three pediatric emergency rulers and all three manikins. The time until each parameter was identified and the value of the parameter were recorded.

Primary outcome was the time needed to identify the four above defined parameters. Secondary outcome was the correctness of the identified parameters and the percentage deviation from the correct value.

ELIGIBILITY:
Inclusion Criteria:

* Medical team members (consultants, residents and nurses) of the department of Anaesthesia at the University Children's Hospital Zurich
* Written informed consent

Exclusion Criteria:

* Having worked with one of the pediatric emergency rulers and knowing where to find the defined parameters

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All medical team members (consultants, residents and nurses) of the department of Anaesthesia at the University Children's Hospital Zurich
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Time to identification | During simulation, approximately 30 minutes
  Time needed to identify the four defined parameters

SECONDARY OUTCOMES:
Correctness | During simulation, approximately 30 minutes
  Correctness of the identified Parameter. The from the participant identified value is compared with the per value defined correctly based on the manikin size.
Percentage deviation | During simulation, approximately 30 minutes
  If the Parameter was identified incorrectly, a percentage deviation of the identified value from the correct value will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Schmidt, MD, Principal Investigator — Department of Anaesthesia and Children's Research Centre, University Children's Hospital, Zurich, Switzerland
Locations (1):
- Department of Anaesthesia and Children's Research Centre, Zurich, Switzerland